CLINICAL TRIAL: NCT04148261
Title: The Effects of Epinephrine and Cortisol on Emotion in Depression
Brief Title: Epinephrine and Cortisol in Depression
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Principal Investigator left lab before study start
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 53325
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — hydrocortisone acetate; Hydrocortisone; epinephrine sulfate; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Arm, CORT + EPI, then PLB + EPI (Active Comparator): Healthy participant will receive cortisol pill and epinephrine infusion
  Interventions: Drug: Hydrocortisone Acetate (CORT); Drug: Epinephrine Sulfate (EPI)
- Healthy Arm, PLB + EPI, then CORT + EPI (Active Comparator): Healthy participant will receive placebo pill and epinephrine infusion
  Interventions: Drug: Epinephrine Sulfate (EPI); Drug: Placebo (PLB)
- Depression Arm, CORT + EPI, then PLB + EPI (Experimental): Depressed participant will receive cortisol pill and epinephrine infusion
  Interventions: Drug: Hydrocortisone Acetate (CORT); Drug: Epinephrine Sulfate (EPI)
- Depression Arm, PLB + EPI, then CORT + EPI (Experimental): Depressed participant will receive placebo pill and epinephrine infusion
  Interventions: Drug: Epinephrine Sulfate (EPI); Drug: Placebo (PLB)

INTERVENTIONS:
Drug: Hydrocortisone Acetate (CORT) — Participants will receive a single dose of hydrocortisone at a dosage of 0.65 mg/kg
  Other Names: Cortef
  Arms: Depression Arm, CORT + EPI, then PLB + EPI; Healthy Arm, CORT + EPI, then PLB + EPI
Drug: Epinephrine Sulfate (EPI) — Participants will receive a continuous infusion of epinephrine at a dosage of 80 ng/kg/min
  Other Names: Adrenalin
Drug: Placebo (PLB) — Participants will receive a placebo
  Arms: Depression Arm, PLB + EPI, then CORT + EPI; Healthy Arm, PLB + EPI, then CORT + EPI

SUMMARY:
This study investigates the effects of two hormones called epinephrine and cortisol on how the brain processes emotional material using functional MRI to measure brain activity. The study hopes to learn how epinephrine and cortisol affect the brain differently in depressed and non-depressed individuals.

ELIGIBILITY:
Inclusion Criteria:

* Weight of less than 280 pounds
* HAM-D Score of greater than 7 for depression participants

Exclusion Criteria:

* Psychotropic medications
* Recent surgery
* Endocrine disorders
* Liver disease
* Kidney disease
* Thyroid disorder
* History of malaria
* Tuberculosis
* Osteoporosis
* Glaucoma or cataracts
* Chronic expressed infections (herpes, HIV, etc)
* History of congestive heart failure
* History of recurring seizures
* Stomach ulcers
* Comorbid psychosis
* Current use of illicit drugs
* Diabetes
* Any cardiovascular disease (angina, hypovolemia, coronary artery disease, low/high blood pressure, etc)
* Any pulmonary disease
* Any cerebrovascular disease
* Sulfate hypersensitivity
* Glaucoma
* Infection
* Pregnancy
* Parkinson's Disease
* Panic Disorder
* Over 280 pounds in weight
* In-dwelling ferrous metals
* Left handed
* Abnormal hearing
* Claustrophobic
* Head injury with loss of consciousness
* Active suicidal ideation

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Sadness-induced subgenual cingulate activity as measured by functional magnetic resonance imaging | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sudheimer, Ph.D., Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No